CLINICAL TRIAL: NCT00236418
Title: Topiramate Clinical Trial in Primary Generalized Tonic-Clonic Seizures
Brief Title: A Study of the Efficacy and Safety of Topiramate in Epilepsy Patients With Primary Generalized Tonic-clonic Seizures
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR005830
Record Dates: First submitted 2005-10-07; First posted 2005-10-12 (Estimated); Last update posted 2011-06-08 (Estimated); Status verified 2010-04

CONDITIONS: Epilepsy; Seizures
Keywords: Epilepsy; Seizures; Topiramate; Prophylaxis; Antiepileptic; Tonic-clonic seizures; Grand mal seizures
MeSH Terms: conditions — Epilepsy; Seizures; Epilepsy, Tonic-Clonic | interventions — Topiramate

INTERVENTIONS:
Drug: topiramate

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of topiramate as an add-on therapy in epilepsy patients with uncontrolled primary generalized tonic-clonic seizures, who are taking 1 or 2 standard antiepileptic drugs.

DETAILED DESCRIPTION:
Epilepsy is a disease characterized by seizures, which are abnormal electrical discharges in the brain that temporarily disrupt normal brain function. Seizures are classified as "generalized," involving all or most of the brain at the same time, or "partial onset," starting in one area of the brain. Generalized tonic-clonic seizures are also referred to as grand mal seizures and are common in people with generalized epilepsy in which the cause is not known. In a tonic-clonic seizure, the person loses consciousness, the body stiffens (tonic phase), and then the individual falls to the ground. This is followed by jerking movements in which the muscles contract and relax quickly (clonic phase). After a minute or two, the jerking movements usually stop, and the person regains consciousness. Antiepileptic medications, such as topiramate, are selected based on a patient's seizure type. Topiramate is a drug that is currently widely used for the treatment of seizures in adults and pediatric patients (2 to 16 years of age). This is a randomized, double-blind, parallel-group, placebo-controlled study to evaluate the effectiveness and safety of topiramate as an add-on therapy in patients with Primary Generalized Tonic-Clonic (PGTC) seizures. The study is in two phases: baseline (8 weeks) and double-blind treatment (20 weeks). Patients are given diaries to record information about their seizures during the phases of the study. During the baseline phase, the patient continues to receive a constant dosage of one or two antiepileptic drugs they have been taking. In the double-blind phase, patients are randomly assigned to either topiramate or placebo. The double-blind phase is divided into two periods: titration, in which the topiramate dose is gradually increased (8 weeks) (patient's antiepileptic medication continues; this dose remains the same) and stabilization (12 weeks). The dose of both topiramate and the patient's antiepileptic drug remain constant during the stabilization period. Based on the investigator's judgment, patients completing the double-blind treatment could enter a long-term extension phase of the study to continue treatment. The primary assessment of effectiveness is the percent reduction in primary generalized tonic-clonic seizure rates from baseline to the double-blind phase. Safety assessments include the frequency of adverse events during the study, results of clinical laboratory tests (hematology, biochemistry, and urinalysis), measurements of vital signs and body weight, physical examination and electrocardiogram (ECG) findings, plasma levels of topiramate and other study antiepileptic drugs, and neurological examinations. The study hypothesis is that topiramate as an add-on is superior to placebo in reducing the seizure rate from baseline to the double-blind phase of the study. Topiramate (25 mg or 100 mg tablets) or placebo, taken by mouth, starting at a dose of 25 or 50mg/day, gradually increasing to a maximum daily dose of 175 mg to 400 mg (based on body weight) or to a maximum tolerated dose (whichever dose is less). Maximum dosage continues for 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Body weight >25 kilograms (55 pounds)
* diagnosis of primary generalized epilepsy
* must have primary generalized tonic-clonic (PGTC) seizures treated with 1 or 2 antiepileptic drugs
* must have three PGTC seizures during baseline period, with at least 1 during each 28-day period of baseline
* females must not have had their first menstrual period or be postmenopausal, or are physically incapable of child bearing, or if of child bearing potential, sexually abstinent, or using adequate birth control measures, and have a negative pregnancy test before study entry.

Exclusion Criteria:

* Patients who do not have epilepsy, such as those with a treatable cause of seizure (for example, active infection or cancer)
* patients with progressive disorders (for example, active infection, cancer or metabolic disturbance)
* patients diagnosed with Lennox-Gastaut syndrome
* history of seizures occurring in only cluster patterns (numerous seizures occurring over a short period of time [<30 minutes])
* documented history (previous 3 months) of generalized tonic-clonic status epilepticus (status epilepticus is a prolonged seizure or seizures repeated frequently over 20 to 30 minutes so that recovery between episodes does not occur) while receiving appropriate antiepileptic medication.

Min Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 1994-12; Study Completion 1996-12 (Actual)

PRIMARY OUTCOMES:
Percent reduction from baseline in primary generalized tonic-clonic seizure rates and percent responders (>=50% reduction in PGTC seizure rate from baseline), during the double-blind phase. Subjects' global evaluation of improvement in seizure severity.

SECONDARY OUTCOMES:
Percent reduction from baseline of all seizure types and percent of treatment responders in all seizure types, during the double-blind phase. Safety evaluations conducted throughout the study.

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- [Result] Montouris GD, Biton V, Rosenfeld WE. Nonfocal generalized tonic-clonic seizures: response during long-term topiramate treatment. Topiramate YTC/YTCE Study Group. Epilepsia. 2000;41(S1):77-81. doi: 10.1111/j.1528-1157.2000.tb02177.x. PMID 10768306
- See also: A study of the efficacy and safety of topiramate in patients with primary generalized tonic-clonic seizures — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=669&filename=CR005830_CSR.pdf